CLINICAL TRIAL: NCT01385644
Title: A Phase I Study to Evaluate the Potential Role of Mesenchymal Stem Cells in the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Evaluate the Potential Role of Mesenchymal Stem Cells in the Treatment of Idiopathic Pulmonary Fibrosis
Acronym: MSC in IPF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Prince Charles Hospital (Other Government)
Collaborators: Mater Medical Research Institute (Other)
Responsible Party: Principal Investigator, Daniel Chambers, Dr Daniel Chambers, The Prince Charles Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC/09/QPCH/105
Record Dates: First submitted 2011-05-04; First posted 2011-06-30 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Mesenchymal stem cells; Idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1*10^6 MSC / kg (Experimental): Placental MSC
  Interventions: Other: Placental MSC
- 2*10^6 MSC / kg (Experimental): Placental MSC
  Interventions: Other: Placental MSC

INTERVENTIONS:
Other: Placental MSC — MSC will be derived from mothers donating their term placenta for clinical trial research purposes at Mater Mothers Hospital, Brisbane. The donation, isolation and expansion of placental-derived MSC for research purposes has been approved by the Mater Health Services (MHS) Human Research Ethics Committee (Reference No. 1292A). These volunteer donor mothers are unrelated to and will be HLA-unmatched with the IPF recipients.

SUMMARY:
The primary objective of this study is to establish the feasibility and safety of infusions of placental Mesenchymal Stem Cells (MSC) from related or unrelated HLA identical or HLA mismatched donors in the treatment of Idiopathic Pulmonary Fibrosis (IPF).

The secondary objectives are to document changes in lung function, 6 minute walk distance (6MWD), gas exchange and radiological appearance following infusion of MSC over a six month evaluation period.

DETAILED DESCRIPTION:
This is a Phase I, open-label, single centre, non-randomized dose-escalation evaluation of the safety and feasibility of MSC treatment for subjects diagnosed with IPF. The first 4 patients will receive a dose of 1 x 10^6 placenta-derived MSC/kg. An interim safety analysis will be carried out by the Data Safety Management Board (DSMB) when these first 4 patients have all undergone their 3 month study visit. Should no serious adverse events be documented due, or likely due, to the MSC infusion, a subsequent 4 patients will receive an IV infusion of 2 x 10^6 placenta-derived MSC/kg. Therefore a total of up to eight (8) subjects who meet all eligibility criteria and who provide written informed consent will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female from 40 to 80 years of age (Note: see exclusion 13 regarding women of child-bearing potential).
2. Diagnosis of IPF based on the following criteria in accordance with American Thoracic Society/European Respiratory Society (ATS-ERS) guidelines for diagnosing

   IPF:

   Definite or probable usual interstitial pneumonia confirmed on surgical lung biopsy (SLB)

   or

   In absence of SLB, all of the following "major criteria"
   * High resolution CT scan (HRCT) showing definite findings for IPF (bibasilar reticular abnormalities with minimal ground glass opacities)
   * Absence of other causes of IPF including drug toxicities, environmental exposure and connective tissue disease
   * Abnormal pulmonary function tests including evidence of a restrictive ventilatory impairment and impaired gas exchange
   * Transbronchial biopsy or BAL suggesting no features of an alternative diagnosis and three of four of the following "minor criteria"
   * Age greater than 50 years
   * Insidious onset of otherwise unexplained dyspnea on exertion
   * Duration of illness greater than 3 months
   * Bibasal, inspiratory crackles

   Within 90 days of study enrolment, diagnosis must be confirmed by HRCT chest.
3. Honeycombing greater than 5% in 0 - 3 lung zones (each lung divided into 3 zones - 1) at the level of the carina 2) highest point of right hemi diaphragm and 3) mid way between these two levels) as assessed on HRCT.
4. Forced vital capacity (FVC) greater than 50 of predicted with a ratio of forced expiratory volume in 1 second to FVC (FEV1/FVC) greater than 0.7 (Pulmonary function tests must be completed no more than 90 days before screening).
5. Diffusing capacity for carbon monoxide (DLCO) greater than 25% of predicted capacity.
6. Ability to perform a 6-Minute Walk Test (6MWT) at screening.
7. Competency to understand the information given in the Human Research and Ethics Committee (HREC) approved ICF and must sign the form prior to the initiation of any study procedures.

Exclusion Criteria:

1. Diagnosis of an interstitial lung disease (ILD) or restrictive lung disease other than IPF.
2. Obstructive lung disease as determined by evidence of airflow obstruction on HRCT or physiologic criteria including:

   FEV1/FVC ratio less than 0.7 Residual volume (RV) greater than 120% by plethysmography or significant (verified by radiologist) emphysema on HRCT if plethysmography not available Evidence of reactive airway disease by change in FEV1 of greater than 12% following bronchodilator challenge
3. Evidence of sustained improvement of IPF condition defined as improvement from pre-therapy pulmonary function tests (PFTs) observed with two or more successive post-therapy PFTs over the year prior to randomization.
4. Active or recent (less than 60 days prior to enrolment) significant respiratory tract infection, or a history of frequent (greater than 2 per year for the last 2 years) infective exacerbations of IPF.
5. Hospitalization within 60 days of screening for an acute exacerbation of IPF (AE-IPF).
6. Chronic heart failure (NYHA class III/IV) or known left ventricular ejection fraction less than 25%.
7. Chronic treatment with the following drugs prescribed for IPF (within 4 weeks of randomization):

   oral corticosteroids (greater than 20 mg/day of prednisone or equivalent), immunosuppressive or cytotoxic drugs, antifibrotic drugs, chronic use of N-acetylcysteine
8. Acute or chronic impairment (other than dyspnea) which limits the ability to comply with study requirements and procedures including the 6MWD
9. Chronic treatment with immunosuppressive, cytotoxic, or antifibrotic drugs including pirfenidone, D-penicillamine, colchicine, cyclosporine A, TNF-alpha antagonists, imatinib, interferon-gamma, cyclophosphamide, or azathioprine within 30 days of randomization.
10. Subject requires hemodialysis, peritoneal dialysis or hemofiltration.
11. Systolic blood pressure less than 85 mmHg.
12. History of malignancies within the past 5 years, with the exception of squamous or basal cell carcinoma of the skin or successfully treated in situ carcinoma of the cervix.
13. Female who is of child-bearing potential.
14. Known history of alcohol abuse within 1 year of enrolment.
15. Participation in a clinical study involving another investigational drug or device within 28 days of screening.
16. Co-morbid condition or illness limiting life expectancy to less than 1 year at time of screening.
17. Serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with treatment, assessment or compliance with the protocol.
18. Significant hypoxemia or hypercapnia at rest on room air as defined by a PaO2 less than 55mmHg or PaCO2 greater than 50mmHg.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chambers, MBBS MRCP FRACP MD, Principal Investigator — The Prince Charles Hospital
Locations (1):
- The Prince Charles Hospital, Brisbane, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All Participants known to doctors through standard of care appointments in clinic.
Pre-assignment Details: All patients meet all inclusion criteria and none of the exclusion criteria.
Period: Overall Study
Arm/Group | 1*10^6 MSC / kg | 2*10^6 MSC / kg
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants meet all inclusion criteria and none of the exclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | 1*10^6 MSC / kg | 2*10^6 MSC / kg | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.1 [62.4 to 66.5] | 66.2 [61.1 to 71.5] | 64.1 [62.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Australia | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Demonstrated Acute Adverse Events Following Infusion
Description: Acute adverse events following infusion was defined as the development of anaphalaxis and/or a 25% increase or decrease from baseline of hemodynamic measurements.
Time Frame: 4 hours post-infusion
Population: Data from 8 participants was analyzed. (4 from each group)
Measure: Number; unit: participants
Arm/Group | 1*10^6 MSC / kg | 2*10^6 MSC / kg
Number analyzed (Participants) | 4 | 4
participants | 0 | 0

2. Secondary Outcome: Percentage Change in Lung Function as Assessed by FVC Compared to Baseline
Description: Forced Vital Capacity (FVC) was measured and reported as a percentage of predicted and comapred from 6 months post-infusion to baseline
Time Frame: 6 months post MSC infusion
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | 1*10^6 MSC / kg | 2*10^6 MSC / kg
Number analyzed (Participants) | 4 | 4
percentage of baseline | 99 [92 to 104] | 94 [90 to 97]

3. Secondary Outcome: Percentage Change in 6 Minute Walk Distance Compared to Baseline
Description: At 6 months 6 Minute Walk Distance was mesured and compared as a percentage to baseline
Time Frame: Baseline and 6 months post MSC infusion
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | 1*10^6 MSC / kg | 2*10^6 MSC / kg
Number analyzed (Participants) | 4 | 4
percentage of baseline | 104 [103 to 114] | 104 [90 to 120]

4. Secondary Outcome: Percentage Change in Lung Function as Assessed by DLCO Compared to Baseline
Description: DLCO was measured as a percentage of predicted, and the percentage change between 6 months post-infusion and baseline is reported.
Time Frame: 6 months post MSC infusion
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | 1*10^6 MSC / kg | 2*10^6 MSC / kg
Number analyzed (Participants) | 4 | 4
percentage of baseline | 117 [96 to 138] | 86 [81 to 96]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the duration of the study participation time which was 12 months.
Arm/Group | 1*10^6 MSC / kg | 2*10^6 MSC / kg
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1*10^6 MSC / kg (N=4) | 2*10^6 MSC / kg (N=4)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient presented with severe abdominal pain. Analgesia, IV antibiotics and hospital admission. CT Scan confirmed small bowel obstruction. Surgery- Small bowel obstruction secondary to band adhesions. Pt recovered and discharged.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1*10^6 MSC / kg (N=4) | 2*10^6 MSC / kg (N=4)
Halitosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) — All pateints experienced halitosis post infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes